CLINICAL TRIAL: NCT05215834
Title: The Comparison of Remimazolam With Propofol in Core Body Temperature in Patients Undergoing Robotic-assisted (RARP) and Laparoscopic (LRP) Radical Prostatectomy
Brief Title: The Comparison of Remimazolam With Propofol in Core Body Temperature
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor, Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: WonkwangUH9
Record Dates: First submitted 2021-12-26; First posted 2022-01-31 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Hypothermia; Anesthesia
Keywords: hypothermia; vasoconstriction threshold; propofol; remimazolam
MeSH Terms: conditions — Hypothermia | interventions — Remifentanil; Propofol; remimazolam

STUDY DESIGN:
Intervention Model Description: Prospective randomized and cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PR group (Active Comparator): Propofol and Remifentanil group
  Interventions: Drug: Remifentanil
- RR group (Experimental): Remimazolam and Remifentanil group
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — 1. Remimazolm and Remifentanil (RR group): anesthesia was induced with remimazolam 6 mg/kg/h by continuous intravenous (IV) infusion and with the effect-site concentration of remifentanil 4 ng/ml and until the loss of consciousness (LoC), followed by remimazolam 1-2 mg/kg/h and remifentanil 3 ng/ml until the end of surgery.
  2. Propofol and Remifentanil (PR group), anesthesia was induced with the effect-site concentration of propofol of 6.0 μg/ml and remifentanil 4 ng/ml, and until the loss of consciousness (LoC), followed by the effect-site concentration of propofol of 2-4 μg/ml and remifentanil 3 ng/ml until the end of surgery.
  Other Names: propofol or remimazolam

SUMMARY:
1. Core body temperature is normally tightly regulated to within a few tenths of a degree. The major thermoregulatory defences in humans are sweating, arteriovenous shunt vasoconstriction, and shivering.
2. Inadvertent hypothermia often complicates prolonged surgery. In patients becoming sufficiently hypothermic, reemergence of thermoregulatory vasoconstriction usually prevents further core hypothermia.
3. The extent to which anesthetics reduce the vasoconstriction threshold depends on the type of drug and its concentration.

DETAILED DESCRIPTION:
1. When propofol induces anesthesia, blood pressure decreases due to vasodilation, which is due to direct action on vascular smooth muscle and vasodilation due to blockage of the sympathetic nervous system. This results in a redistribution of body temperature, resulting in hypothermia.
2. The effects of remimazolam on the central nervous system, respiratory and cardiovascular system have been studied. Remimazolam, a new type of benzodiazepine drug acts on the GABA-A receptor and has the advantages of rapid induction, rapid recovery, stable hemodynamics, and mild respiratory inhibition. At present, there is little literature on its practice in intraoperative thermoregulation under general anesthesia.
3. Investigators hypothesized that the type of anesthetic agents might affect thermoregulatory mechanisms such as the redistribution of body heat, cutaneous heat loss or inhibition of thermoregulatory vasoconstriction. Therefore, Investigators investigated to compare remimazolam with propofol in core body temperature, vasoconstriction threshold and times to onset of vasoconstriction(min)in patients given laparoscopic assisted vaginal hysterectormy.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical classification I-III,
2. Patients who undergoing Robotic-assisted or laparoscopic (LRP) radical prostatectomy.

Exclusion Criteria:

1. Patients who have Medications or any implanted device that could affect cardiovascular function
2. Patients who have a history with heat imbalance, thyroid diseases, dystautonomia, Raynaud's syndrome, uncontrolled diabetes mellitus, or hypertension.

Ages: 19 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
core body temperature change (°C) | at 60 minutes after induction of general anesthesia
  After the induction of general anesthesia, a nasopharyngeal temperature probe was inserted through the nasal cavity, and a 9.5- to 10.0-cm depth was set for optimal placement. The nasopharyngeal temperature was recorded every 10 min until the end of surgery

SECONDARY OUTCOMES:
times to onset of vasoconstriction (minute) | From after induction to until the end of surgery
  time to arrive the skin temperature gradient (between forearm and index finger tip) equaled 0 °C.
intraoperative hypothermia | From after induction to until the end of surgery
  core body temperature of <36 °C in patients undergoing anesthesia and surgery
Mean arterial pressure (mmHg) | From after induction to until the end of surgery
  Mean arterial pressure
Heart rate (beats/min) | From after induction to until the end of surgery
  Heart rate
vasoconstriction threshold (°C) | From after induction to until the end of surgery
  the tympanic membrane temperature at which the skin temperature gradient (between forearm and index finger tip) equaled 0 °C

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Lee, M.D.,Ph.D, Principal Investigator — Department of anesthesiology and pain medicine, Wonkwang University Hospital
Locations (1):
- Wonkwag UH, Iksan, South Korea